CLINICAL TRIAL: NCT02662114
Title: A European Multi-centre, Retrospective, Non-interventional Study of the Effectiveness of Tresiba® (Insulin Degludec) After Switching Basal Insulin in a Population With Type 1 or Type 2 Diabetes Mellitus
Brief Title: Investigating the Effectiveness of Tresiba® (Insulin Degludec) After Switching Basal Insulin in a Population With Type 1 or Type 2 Diabetes Mellitus
Acronym: EU-TREAT
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1250-4240; U1111-1170-3128 (Other: WHO)
Record Dates: First submitted 2015-12-04; First posted 2016-01-25 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tresiba®
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Information will be collected from the medical records (paper/electronic) of each patient at several outpatient clinics to describe the two periods of medical history: before and after the initiation date of Tresiba®. For each patient, data will be collected, to describe a minimum of 6 months to a maximum of 12 months in each period; thus, the study will collect information on 12 to 24 months of medical history for each patient.

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the effectiveness of Tresiba® (insulin degludec) after switching basal insulin in a population with type 1 or type 2 diabetes mellitus.

EU-TREAT (EUropean TREsiba AudiT)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained before any study-related activities. Study-related activities are any data collection from the medical records of the patient
* Age at least 18 years at the time of Tresiba® initiation
* T1DM or insulin-treated T2DM patients
* Switched to Tresiba® (with or without prandial insulin) after any basal insulin (with or without prandial insulin). Switch must have occurred at least 6 months prior to data collection and the patient may or may not be treated with Tresiba® at the time of patient selection
* Previously treated with any basal insulin (with or without prandial insulin) for at least 6 months prior to switching to Tresiba®
* At least one documented medical visit in the first 9 months after Tresiba® initiation
* Minimum available data at the time of Tresiba® initiation: age, type of diabetes, HbA1c (Glycated haemoglobin), duration of diabetes, duration and type of insulin treatment, medical follow-up at the study site of at least 1 year, and an eGFR (Estimated glomerular filtration rate )value in the last 12 months

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having signed the Informed Consent
* Participation in a diabetes clinical trial or receipt of any investigational medicinal product up to 12 months before or any time after the initiation of Tresiba®
* Current participation in another non-interventional study on insulin degludec (Tresiba®)
* Patients treated by continuous subcutaneous insulin infusion or premix insulin in the 6 months prior to receiving Tresiba®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T1DM (Type 1 diabetes mellitus) and T2DM (Type 2 diabetes mellitus) patient sample treated with Tresiba® under conditions of routine care.
Sampling Method: Non-Probability Sample
Enrollment: 2302 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2016-08-12 (Actual); Study Completion 2016-08-12 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c after switch to Tresiba® | Month 0, Month 6

SECONDARY OUTCOMES:
Change in HbA1c after switch to Tresiba® | Month 0, Month 12
Change in the percentage of patients with HbA1c below recommended targets (below 7.0%, 7.5%, and 8.0%) after switch to Tresiba® | Month 0, Month 6
Change in the percentage of patients with HbA1c below recommended targets (below 7.0%, 7.5%, and 8.0%) after switch to Tresiba® | Month 0, Month 12
Change in the mean FPG (Fasting Plasma Glucose ) level after switch to Tresiba® | Month 0, Month 6
Change in the mean FPG level after switch to Tresiba® | Month 0, Month 12
Tresiba® starting dose at switch and doses | At 6 months
Tresiba® starting dose at switch and doses | At 12 months
Change in the mean daily insulin doses (total, basal, prandial) after switch to Tresiba® | Month 0, Month 6
Change in the mean daily insulin doses (total, basal, prandial) after switch to Tresiba® | Month 0, Month 12
Change in the number of concomitant non-insulin glucose-lowering drug classes after switch to Tresiba® | Month 0, Month 6
Change in mean dose of concomitant non-insulin glucose-lowering drug classes after switch to Tresiba® | Month 0, Month 6
Change in the number of concomitant non-insulin glucose-lowering drug classes after switch to Tresiba® | Month 0, Month 12
Change in mean dose of concomitant non-insulin glucose-lowering drug classes after switch to Tresiba® | Month 0, Month 12
Change in body weight (kg) after switch to Tresiba® | Month 0, Month 6
Change in body weight (kg) after switch to Tresiba® | Month 0, Month 12
Change in the percentage of patients with at least one hypoglycaemic episode (overall, non-severe, severe, nocturnal) before and after switch to Tresiba® | -6 to 0 months ie 6 months before switch to Tresiba®
Change in the percentage of patients with at least one hypoglycaemic episode (overall, non-severe, severe, nocturnal) before and after switch to Tresiba® | 0 to +6 months
Change in the percentage of patients with at least one hypoglycaemic episode (overall, non-severe, severe, nocturnal) before and after switch to Tresiba® | -12 to 0 months ie 12 months before switch to Tresiba®
Change in the percentage of patients with at least one hypoglycaemic episode (overall, non-severe, severe, nocturnal) before and after switch to Tresiba® | 0 to +12 months
Change in the rates of hypoglycaemic episodes (overall, non-severe, severe, nocturnal) before and after switch to Tresiba® (per patient-month) | -6 to 0 months ie 6 months before switch to Tresiba®
Change in the rates of hypoglycaemic episodes (overall, non-severe, severe, nocturnal) before and after switch to Tresiba® (per patient-month) | 0 to +6 months
Change in the rates of hypoglycaemic episodes (overall, non-severe, severe, nocturnal) before and after switch to Tresiba® (per patient-month) | -12 to 0 months ie 12 months before switch to Tresiba®
Change in the rates of hypoglycaemic episodes (overall, non-severe, severe, nocturnal) before and after switch to Tresiba® (per patient-month) | 0 to +12 months
Change in the number of ER (Emergency Room) visits related to hypoglycaemia after switch to Tresiba® | -6 to 0 months ie 6 months before switch to Tresiba®
Change in the number of ER visits related to hypoglycaemia after switch to Tresiba® | 0 to +6 months
Change in the number of ER visits related to hypoglycaemia after switch to Tresiba® | -12 to 0 months ie 12 months before switch to Tresiba®
Change in the number of ER visits related to hypoglycaemia after switch to Tresiba® | 0 to +12 months
Change in the number of HCP (Healthcare professional(s)) visits related to hypoglycaemia after switch to Tresiba® | -6 to 0 months (ie 6 months before switch to Tresiba®)
Change in the number of HCP visits related to hypoglycaemia after switch to Tresiba® | 0 to +6 months
Change in the number of HCP visits related to hypoglycaemia after switch to Tresiba® | -12 to 0 months ie 12 months before switch to Tresiba®
Change in the number of HCP visits related to hypoglycaemia after switch to Tresiba® | 0 to +12 months
Change in the number of hospitalisations related to hypoglycaemia after switch to Tresiba® | -6 to 0 months ie 6 months before switch to Tresiba®
Change in the number of hospitalisations related to hypoglycaemia after switch to Tresiba® | 0 to +6 months
Change in the number of hospitalisations related to hypoglycaemia after switch to Tresiba® | -12 to 0 months ie 12 months before switch to Tresiba®
Change in the number of hospitalisations related to hypoglycaemia after switch to Tresiba® | 0 to +12 months
Percentage of patients continuing Tresiba® post-switch | At 6 months
Percentage of patients continuing Tresiba® post-switch | At 12 months
Reason(s) for starting Tresiba®, if available | Month 0, Month 12
Reason(s) for discontinuing Tresiba®, if applicable and available | Month 0, Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (6):
- Novo Nordisk Investigational Site, Vienna, Austria
- Novo Nordisk Investigational Site, Gentofte Municipality, Denmark
- Novo Nordisk Investigational Site, München, Germany
- Novo Nordisk Investigational Site, Athens, Greece
- Novo Nordisk Investigational Site, Perugia, Italy
- Novo Nordisk Investigational Site, Sankt Gallen, Switzerland

REFERENCES:
- [Result] Siegmund T, Tentolouris N, Knudsen ST, Lapolla A, Prager R, Phan TM, Wolden ML, Schultes B; EU-TREAT study group. A European, multicentre, retrospective, non-interventional study (EU-TREAT) of the effectiveness of insulin degludec after switching basal insulin in a population with type 1 or type 2 diabetes. Diabetes Obes Metab. 2018 Mar;20(3):689-697. doi: 10.1111/dom.13149. Epub 2017 Nov 21. PMID 29106039
- [Result] Tentolouris N, Knudsen ST, Lapolla A, Wolden ML, Haldrup S, Schultes B. Switching "Real-World" Diabetes Patients to Degludec from Other Basal Insulins Provides Different Clinical Benefits According to Their Baseline Glycemic Control. Adv Ther. 2019 May;36(5):1201-1210. doi: 10.1007/s12325-019-00916-7. Epub 2019 Mar 16. PMID 30879256
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com